CLINICAL TRIAL: NCT04173442
Title: Post-Authorization Safety Study to Monitor Pregnancy and Infant Outcomes Following Administration of Dupilumab During Planned or Unexpected Pregnancy in North America
Brief Title: Post-authorization Safety Study in North America to Monitor Pregnancy and Infant Outcomes Following Administration of Dupilumab During Planned or Unexpected Pregnancy
Status: Recruiting | Type: Observational
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: R668-AD-1639
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Atopic Dermatitis (AD); Asthma
MeSH Terms: conditions — Dermatitis, Atopic; Asthma | interventions — dupilumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: Dupilumab-Exposed Cohort: Pregnant women with approved indications exposed to dupilumab during pregnancy
  Interventions: Drug: dupilumab
- Cohort 2: Disease-Matched Comparison Cohort: Pregnant women with approved indications not exposed to dupilumab during pregnancy
- Cohort 3: Healthy Comparison Cohort: Pregnant women who are not diagnosed with any dupilumab-approved indications, and not exposed to dupilumab during pregnancy

INTERVENTIONS:
Drug: dupilumab — Dupilumab cohort
  Other Names: REGN668; Dupixent®; SAR23189
  Groups: Cohort 1: Dupilumab-Exposed Cohort

SUMMARY:
The objective is to evaluate the potential effect of exposure to dupilumab in pregnancy compared to the primary comparison group of disease-matched pregnant women who are not exposed to dupilumab, and the secondary comparison group of healthy pregnant women.

The primary outcome of the study is major structural defects, and the secondary outcomes of the study are spontaneous abortion/miscarriage, stillbirth, elective termination/abortion, premature delivery, small for gestational age, pattern of 3 or more minor structural defects, postnatal growth of live born children to 1 year of age, postnatal serious or opportunistic infections in live born children to 1 year of age, and hospitalizations in live children up to 1 year of age.

ELIGIBILITY:
Key Inclusion Criteria:

Cohort 1: Dupilumab-Exposed Cohort

* Pregnant women
* Exposure to dupilumab for the treatment of the approved indications of atopic dermatitis (AD) or asthma, for any number of days, at any dose, and at any time from the first day of the LMP up to and including the end of pregnancy.

Cohort 2: Disease-Matched Comparison Cohort (Comparison Group 1)

* Pregnant women
* Diagnosed with a dupilumab-approved indications of moderate-to-severe AD without asthma or moderate-to-severe asthma; frequency matched to the exposed group by disease indication, with the indication and severity validated by medical records when possible.
* No exposure to dupilumab any time in the current pregnancy or within 10 weeks of the first day of the LMP and may or may not have taken another medication for their disease in the current pregnancy.

Cohort 3: Healthy Comparison Cohort (Comparison Group 2):

* Pregnant women

Key Exclusion Criteria:

Cohort 1: Dupilumab-Exposed Cohort

* Women who have first contact with the project after prenatal diagnosis of any major structural defect
* Women who have used dupilumab for an indication other than asthma or AD

Cohort 2: Disease-Matched Comparison Cohort (Comparison Group 1):

* Women who have first contact with the project after prenatal diagnosis of any major structural defect
* Exposure to dupilumab within 10 weeks of LMP or anytime during the current pregnancy

Cohort 3: Non-Diseased Comparison Cohort (Comparison Group 2):

* Exposure to dupilumab within 10 weeks prior to the first day of the LMP
* Women who have a diagnosis of any dupilumab approved indication
* Women who have first contact with the project after prenatal diagnosis of any major structural defect

NOTE: Other protocol defined Inclusion/Exclusion Criteria apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study population includes pregnant women who reside in the US or Canada with dupilumab- exposure for the approved indication, and 2 comparison groups without dupilumab exposure during pregnancy (1 disease-matched unexposed comparison group, and 1 healthy unexposed comparison group).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-10-24 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Rate of major structural defects | Up to 1 Year of Age
  Defined and classified using the Centers for Disease Control and Prevention (CDC) coding manual that is used for the Metropolitan Atlanta Congenital Defects Program (MACDP) classification of major structural defects

SECONDARY OUTCOMES:
Incidence of spontaneous abortion or miscarriage | Up to 20 weeks post-LMP (Last Menstrual period)
  Defined as non-deliberate fetal death
Incidence of stillbirth | At or after 20 weeks post-LMP
  Defined as non-deliberate fetal death
Incidence of elective termination/abortion | Up to 9 months
  Defined as deliberate discontinuation of pregnancy through medication or surgical procedures
Incidence of premature delivery | Prior to 37 weeks of gestation
  Defined as live birth prior to 37.0 weeks gestation as counted from LMP (or ultrasound-adjusted date)
Incidence of small for gestational age | At Birth
  Defined as birth size (weight, length or head circumference) less than or equal to the 10th centile for sex and gestational age using standard pediatric CDC growth curves for full term or preterm infants
Incidence of a pattern of 3 or more minor structural defects | Between Birth and Up to 1 Year of Age
  Identified by a study examiner: Defined as 1 of the defects representing a structural anomaly which has neither cosmetic nor functional significance to the child
Postnatal growth deficiency | Up to 1 Year of Age
  Defined as postnatal size (weight, length or head circumference) less than or equal to the 10th centile for sex and age using standard pediatric growth curves, and adjusted for postnatal age for premature infants if the postnatal measurement is obtained at less than 1 year of age.
Incidence of postnatal serious or opportunistic infections in live born children | Up to 1 Year of Age
  Defined as any infection resulting in hospitalization
Incidence of hospitalizations in live born children | Up to 1 Year of Age
  Defined as any hospitalization of the infant within the first year of life after discharge following delivery

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Regeneron Research Site, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No